CLINICAL TRIAL: NCT03682575
Title: Work of Breathing and Oxygen Saturation Stability in Premature Infants With History of Respiratory Insufficiency Prior to Discharge
Brief Title: Work of Breathing in Premature Infants at Discharge
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: DDD604122
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Bronchopulmonary Dysplasia; Very Low Birth Weight Infant; Prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants WITH diagnosis of bronchopulmonary dysplasia (BPD): Preterm infants who were on oxygen at 28 days of life.
  Interventions: Other: Enrollment
- Infants WITHOUT diagnosis of bronchopulmonary dysplasia (BPD: Preterm infants who were not on oxygen at 28 days of life.
  Interventions: Other: Enrollment

INTERVENTIONS:
Other: Enrollment — All infants whose families consent will be enrolled and will all receive the same treatment which included measurements of work of breathing.

SUMMARY:
The purpose of this study is to compare how premature infants who required oxygen for at least 28 days during their time in the NICU (Neonatal Intensive Care Unit) breathe at discharge compared to premature infants who did not require oxygen for at least 28 days during their time in the NICU.

DETAILED DESCRIPTION:
Work of breathing tests will be performed on premature infants who required oxygen for at least 28 days during their time in NICU. These same work of breathing tests will be performed in another group of premature infants who did not require oxygen for at least 28 days during their time in the NICU. The two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at greater than 26 weeks gestation, weighing less than 1500 grams at birth.
* Infants with diagnosis of BPD and without diagnosis of BPD

Exclusion Criteria:

* Infants with skeletal, neuromuscular, or abdominal surgical disorders that affect the accuracy of work of breathing measurements will be excluded.

Ages: 1 Month to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants born greater than 26 weeks gestation, weighing less than 1500 grams at birth. Work of breathing indices will be compared between the group of babies who were diagnosed with BPD and the group that was not diagnosed with BPD.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Work of breathing indices | 25 minutes
  Respiratory Inductance Plethysmography (RIP) measurements will be taken and Phase Angle will be measured.

SECONDARY OUTCOMES:
Intermittent Hypoxia | 25 minutes
  Oxygen saturation will be measured using a high resolution pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Z Kovatis, MD, Principal Investigator — ChristianaCare
Locations (1):
- Christiana Care Health Services, Inc, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No